CLINICAL TRIAL: NCT00449293
Title: Behavioral Therapy for Reduction in Smoking Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0606054
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2008-01

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: Smoking cessation; Tobacco dependence; Mindfulness; fMRI; Craving
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: standard cognitive behavioral therapy
- 2 (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy

INTERVENTIONS:
Behavioral: standard cognitive behavioral therapy — Standard therapy to help participants with smoking cessation.
  Arms: 1
Behavioral: Mindfulness Based Cognitive Therapy — A novel mind body therapy that extends basic CT principles to include the practice of mindfulness, which fosters a dispassionate approach to the experience of craving.
  Arms: 2

SUMMARY:
The objective of this pilot research is to investigate the effects of two behavioral smoking cessation programs on aspects of cue-induced cigarette craving, and to further investigate the neural bases of such effects.

DETAILED DESCRIPTION:
The objective of this pilot research is to investigate the effects of two behavioral smoking cessation programs on aspects of cue-induced cigarette craving, and to further investigate the neural bases of such effects. The specific objectives of the study include 1) to investigate the effects of behavioral therapy on cue induced craving using a cognitive task and a fMRI paradigm 2) to pilot test questionnaires and study procedures, and 3) to gather preliminary estimates of the effect size of the novel behavioral therapy for smoking cessation in order to inform the design of a larger trial. A secondary goal of this research is 1) to determine the impact of two cognitive coping techniques on attentional bias to smoking related cues as measured by behavioral responses and patterns of neural activation and 2) to determine the impact of two cognitive coping techniques on cue-induced cigarette craving as measured by self-report and patterns of neural activation. Daily smokers desiring to quit smoking were randomized to one of two behavioral smoking cessation programs: (1) standard cognitive behavioral therapy or (2) mindfulness-based cognitive therapy. Participants completed questionnaires and a brief computer-based cognitive testing paradigm. Participants also underwent a fMRI scan at quit day (week 5). A randomly assigned subset of the participants (n= 18), underwent two additional scans at baseline (week 1) and end-of-therapy (week 8). The study has thus used self-report measures, cognitive testing (Stroop task), and fMRI (functional magnetic resonance imaging) assessments.

ELIGIBILITY:
Inclusion Criteria:

* Currently be cigarette smokers who desire to quit in the next 30 days (preparation phase).
* Subjects must smoke at least 10 cigarettes per day
* Must be at least 18 years old
* English speaking
* Able to read, understand, and complete a written questionnaire
* Must be willing to attend 8 sessions of behavioral therapy and perform daily home practice
* Must not currently be using pharmacologic therapy to quit
* Must also be willing to abstain from pharmacologic therapy for the duration of the study, which is 8 weeks from the time of enrollment.
* Only strongly right-handed subjects will be included

Exclusion Criteria:

* Pregnant women
* Have metal permanently in or on the body (aneurysm clips, permanent piercings, permanent dental work)
* Weigh over 300 pounds
* Known problem of claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention of participants | baseline - session 8 and 6 month follow-up
Participant acceptability of novel behavioral intervention (mindfulness) | baseline - session 8

SECONDARY OUTCOMES:
Smoking cessation | baseline - session 8 and 6 month follow-up
Exhaled CO readings | baseline, sessions 5 & 8
Salivary cotinine measures | baseline and sessions 5 & 8
Psychological Measures | baseline & session 8
Craving response from a smoking cue (fMRI) | Sessions 1,5, & 8
Reaction times on Smoking Stroop tasks (behavioral and fMRI-administered) | Sessions 1,5, & 8
Self Reported Measures: | baseline, sessions 5 & 8
Trait Self-Control Scale | baseline & session 8
State Ego Depletion Scale | baseline & session 8
Self-Efficacy Scale | baseline & session 8
Perceived Stress Scale | baseline & session 8
Positive and Negative Affect Scale | baseline & session 8
Difficulties in Emotional Regulation Scale | baseline & session 8
Snaith-Hamilton Hedonic Capacity Scale | baseline & session 8
Mindful Attention Awareness Scale | baseline & session 8
Kentucky Inventory of Mindfulness Scales | baseline & session 8
Mindfulness meditation practice (mindfulness participants only, time in minutes | sessions 1-8

CONTACTS AND LOCATIONS:
Overall Officials: Hilary A Tindle, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Astin JA, Shapiro SL, Eisenberg DM, Forys KL. Mind-body medicine: state of the science, implications for practice. J Am Board Fam Pract. 2003 Mar-Apr;16(2):131-47. doi: 10.3122/jabfm.16.2.131. PMID 12665179
- [Background] Baer RA, Smith GT, Allen KB. Assessment of mindfulness by self-report: the Kentucky inventory of mindfulness skills. Assessment. 2004 Sep;11(3):191-206. doi: 10.1177/1073191104268029. PMID 15358875
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Gilbert DG, McClernon FJ, Rabinovich NE, Dibb WD, Plath LC, Hiyane S, Jensen RA, Meliska CJ, Estes SL, Gehlbach BA. EEG, physiology, and task-related mood fail to resolve across 31 days of smoking abstinence: relations to depressive traits, nicotine exposure, and dependence. Exp Clin Psychopharmacol. 1999 Nov;7(4):427-43. doi: 10.1037//1064-1297.7.4.427. PMID 10609977
- [Background] Speca M, Carlson LE, Goodey E, Angen M. A randomized, wait-list controlled clinical trial: the effect of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients. Psychosom Med. 2000 Sep-Oct;62(5):613-22. doi: 10.1097/00006842-200009000-00004. PMID 11020090